CLINICAL TRIAL: NCT03255109
Title: WEAN SAFE (WorldwidE AssessmeNt of Separation of pAtients From Ventilatory assistancE)
Brief Title: WorldwidE AssessmeNt of Separation of pAtients From Ventilatory assistancE
Acronym: WEAN SAFE
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: WEAN SAFE
Record Dates: First submitted 2017-08-09; First posted 2017-08-21 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Acute Severe Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Lung; acute; respiratory; distress; weaning; mechanical ventilation; respiratory infection
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
WEAN SAFE (WorldwidE AssessmeNt of Separation of pAtients From ventilatory assistancE) is a multi-centre, prospective, observational, 4-week inception cohort study being carried out by the Acute Respiratory Failure section of ESICM. Weaning represents a challenge for intensivists and patients spend a considerable amount of time in being liberated from mechanical ventilation. While guidelines do exist on the classification of weaning, a recent study has shown that these may not be applicable to all patients. Moreover, different practices exist in regard to weaning procedures. WEAN SAFE will prospectively assess the burden of, management and spectrum of approaches to weaning from ventilation, in patients that require invasive mechanical ventilation for any reason, for a time period of at least 24 hours.

DETAILED DESCRIPTION:
The purpose of this study is to describe, in a large population of ICU patients the burden of, management and spectrum of approaches to weaning from ventilation, in patients that require invasive mechanical ventilation for any reason, for a time period of at least 24 hours. It will answer the following questions:

* What are the current approaches taken to wean patients from invasive mechanical ventilation?
* What is the frequency of delayed weaning from invasive mechanical ventilation?
* What are the factors that are used to determine when patients are in the weaning phase?
* What are the barriers to effective weaning from invasive MV?
* What factors (patient, institutional, medical practice) contribute to failed attempts to wean from invasive mechanical ventilation?
* What is the impact of premorbid conditions on weaning from invasive MV?
* What is the utility of existing classifications for weaning from invasive MV?
* What is the impact of early versus delayed and/or failed weaning from invasive MV?

Patients will be screened for the study when undergoing mechanical ventilation and admitted in the ICU.

Day 1 will be defined as the first day when IMV commences Day 2 commences at 6-10am (fixed time point each day per ICU practice) after IMV commences. Patients undergoing invasive mechanical ventilation on the morning of day 1 will be screened for the study Patients still undergoing IMV on Day 2, will be enrolled in the study Patients not undergoing invasive mechanical ventilation or liberated from invasive mechanical ventilation on day 1 will be re-evaluated daily for the presence of inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

Screening: all patients admitted in the ICU and aged >16 will be screened daily

- A patient will be included if he/she is undergoing Invasive mechanical ventilation on the second morning (between 6am and 10 am) after initiation of mechanical ventilation or after ICU admission (if ventilation was already in place).

Exclusion Criteria:

* Lack of informed consent (where required)
* Patients already present in the ICU at the beginning of the study, independently of the form of ventilatory support

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Due to the observational nature of the present study, patients enrolled in other observational/interventional study CAN be enrolled in the present study.
  We aim to collect a large "convenience sample", with > 5,000 patients. Based on the LUNG SAFE data (NCT02010073; JAMA, 2016 Jul 19;316(3):347), we can estimate to enroll about 11 patients invasively ventilated on Day 2 following intubation per participating ICU in a 4 week period. We are therefore targeting the enrollment of 500 registered ICUs (considering a 10% dropout)
Sampling Method: Probability Sample
Enrollment: 11000 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The number of patients invasively ventilated in the last 24 hours | 90 days or hospital discharge (whichever occurs first)
  To describe the frequency of simple, difficult and prolonged weaning

SECONDARY OUTCOMES:
The current approaches taken to wean patients from invasive mechanical ventilation and impact on weaning duration | 90 days or hospital discharge (whichever occurs first)
  What are the factors ((patient, institutional, medical practice) that are used to determine when patients are in the weaning phase

CONTACTS AND LOCATIONS:
Overall Officials: John LAFFEY, MD, Principal Investigator — National University of Galway, Ireland and St Michael's Hospital-University of Toronto, Canada; Giacomo BELLANI, MD, Principal Investigator — S Gerardo Hospital, University of Milan-Bicocca, Monza, Italy
Locations (1):
- All Centres From All Over the World Willing to Contribute Are Welcome, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Background] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Background] Fagon JY, Chastre J, Vuagnat A, Trouillet JL, Novara A, Gibert C. Nosocomial pneumonia and mortality among patients in intensive care units. JAMA. 1996 Mar 20;275(11):866-9. PMID 8596225
- [Background] Epstein SK, Ciubotaru RL. Independent effects of etiology of failure and time to reintubation on outcome for patients failing extubation. Am J Respir Crit Care Med. 1998 Aug;158(2):489-93. doi: 10.1164/ajrccm.158.2.9711045. PMID 9700126
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924
- [Background] Blackwood B, Alderdice F, Burns K, Cardwell C, Lavery G, O'Halloran P. Use of weaning protocols for reducing duration of mechanical ventilation in critically ill adult patients: Cochrane systematic review and meta-analysis. BMJ. 2011 Jan 13;342:c7237. doi: 10.1136/bmj.c7237. PMID 21233157
- [Background] Ely EW, Baker AM, Dunagan DP, Burke HL, Smith AC, Kelly PT, Johnson MM, Browder RW, Bowton DL, Haponik EF. Effect on the duration of mechanical ventilation of identifying patients capable of breathing spontaneously. N Engl J Med. 1996 Dec 19;335(25):1864-9. doi: 10.1056/NEJM199612193352502. PMID 8948561
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Beduneau G, Pham T, Schortgen F, Piquilloud L, Zogheib E, Jonas M, Grelon F, Runge I, Nicolas Terzi, Grange S, Barberet G, Guitard PG, Frat JP, Constan A, Chretien JM, Mancebo J, Mercat A, Richard JM, Brochard L; WIND (Weaning according to a New Definition) Study Group and the REVA (Reseau Europeen de Recherche en Ventilation Artificielle) Network double dagger. Epidemiology of Weaning Outcome according to a New Definition. The WIND Study. Am J Respir Crit Care Med. 2017 Mar 15;195(6):772-783. doi: 10.1164/rccm.201602-0320OC. PMID 27626706
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Derived] Pham T, Heunks L, Bellani G, Madotto F, Aragao I, Beduneau G, Goligher EC, Grasselli G, Laake JH, Mancebo J, Penuelas O, Piquilloud L, Pesenti A, Wunsch H, van Haren F, Brochard L, Laffey JG; WEAN SAFE Investigators. Weaning from mechanical ventilation in intensive care units across 50 countries (WEAN SAFE): a multicentre, prospective, observational cohort study. Lancet Respir Med. 2023 May;11(5):465-476. doi: 10.1016/S2213-2600(22)00449-0. Epub 2023 Jan 21. PMID 36693401
- See also: webpage on Wean Safe where more useful details can be found such as the link to register your site — http://www.esicm.org/research/WEAN-SAFE